CLINICAL TRIAL: NCT07024797
Title: A Multiple Ascending Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of ABBV-932 in Healthy Adult Chinese Subjects
Brief Title: Study to Assess the Adverse Events, Tolerability, and How Oral Doses of ABBV-932 Moves Through the Body in Healthy Adult Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M25-644
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-932

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ABBV-932 or Placebo Part A (Experimental): Participants will receive oral ABBV-932 or placebo once daily (QD) for 14 days.
  Interventions: Drug: ABBV-932; Drug: Placebo for ABBV-932
- ABBV-932 or Placebo Part B (Experimental): Participants will receive oral ABBV-932 or placebo QD for 14 days.
  Interventions: Drug: ABBV-932; Drug: Placebo for ABBV-932
- ABBV-932 or Placebo Part C (Experimental): Participants will receive oral ABBV-932 or placebo QD 42 days.
  Interventions: Drug: ABBV-932; Drug: Placebo for ABBV-932

INTERVENTIONS:
Drug: ABBV-932 — Oral Capsule
Drug: Placebo for ABBV-932 — Oral Capsule

SUMMARY:
This study will assess the adverse events, tolerability, and how oral doses of ABBV-932 moves through the body in healthy adult Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 to ≤ 27.9 kg/m^2 after rounding to the tenths decimal. BMI is calculated as weight in kg divided by the square of height measured in meters.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, unexplained syncope, or any uncontrolled medical illness.
* History of suicidal ideation within one year prior to study treatment administration as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the C-SSRS completed at Screening, or any history of suicide attempts as evidenced by answering "yes" to any suicidal behavior question (except a "yes" to the "Has subject engaged in non-suicidal self-injurious behavior" question) within the last 2 years.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-08-21 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ABBV-932 | Up to approximately 43 days
  Cmax of ABBV-932
Time to Cmax (Tmax) of ABBV-932 | Up to approximately 43 days
  Tmax of ABBV-932
Observed plasma concentration at the end of a dosing interval (Ctrough) of ABBV-932 | Up to approximately 43 days
  Ctrough of ABBV-932
Area under the plasma concentration-time curve from time 0 until the last measurable concentration (AUCtau) of Desmethyl Cariprazine ABBV-932 | Up to approximately 43 days
  AUCtau of ABBV-932
Maximum Plasma Concentration (Cmax) of DCAR | Up to approximately 43 days
  Cmax of DCAR
Time to Cmax (Tmax) of DCAR | Up to approximately 43 days
  Tmax of DCAR
Observed plasma concentration at the end of a dosing interval (Ctrough) of DCAR | Up to approximately 43 days
  Ctrough of DCAR
Area under the plasma concentration-time curve from time 0 until the last measurable concentration (AUCtau) of Desmethyl Cariprazine (DCAR) | Up to approximately 43 days
  AUCtau of DCAR
Maximum Plasma Concentration (Cmax) of Didesmethyl-Cariprazine (DDCAR) | Up to approximately 43 days
  Cmax of DDCAR
Time to Cmax (Tmax) of DDCAR | Up to approximately 43 days
  Tmax of DDCAR
Observed plasma concentration at the end of a dosing interval (Ctrough) of DDCAR | Up to approximately 43 days
  Ctrough of DDCAR
Area under the plasma concentration-time curve from time 0 until the last measurable concentration (AUCtau) of DDCAR | Up to approximately 43 days
  AUCtau of DDCAR
Number of Participants Experiencing Adverse Events | Up to approximately 75 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Shanghai Mental Health Center /ID# 273427, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-644